CLINICAL TRIAL: NCT06463782
Title: Phase I Clinical Trial of the Safety, Pharmacokinetics, Biodistribution and Dosimetry of 68Ga-LNC1007 Injection in Adult Healthy Volunteers and Solid Tumor Patients
Brief Title: Clinical Study of 68Ga-LNC1007 Injection PET/CT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yantai LNC Biotechnology Singapore PTE. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 68Ga-LNC1007-001
Record Dates: First submitted 2024-06-04; First posted 2024-06-18 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers; Cancer Patients

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 68Ga-LNC1007 Injection (Experimental): a single dose of 68Ga-LNC1007 Injection will be administered
  Interventions: Drug: 68Ga-LNC1007 Injection

INTERVENTIONS:
Drug: 68Ga-LNC1007 Injection — The participant will receive a single intravenous injection with 0.05 mCi/kg (according to the participants' body weight) 68Ga-LNC1007 Injection on the scan bed. The final dose of the drug is allowed to fluctuate within the 20% range, but not below 3 mCi. A 10 mL normal saline flush will be given after the completion of the injection to ensure the residue is injected.

SUMMARY:
This study is a single-arm, single-center trial aimed at evaluating the safety, pharmacokinetics, biodistribution and dosimetry of 68Ga-LNC1007 Injection in adult healthy volunteers and solid tumor patients.

All participants must provide a signed informed consent form before enrolling in the trial.

A total of 8 adult healthy volunteers and solid tumor patients will be involved in the trial. There should be no less than 3 and no more than 5 participants in either group. If any participant drops out during the trial, or an effective scan image becomes unavailable, additional volunteers will be recruited to ensure the sample size. The participant will receive a single intravenous injection with 68Ga-LNC1007 Injection.Each subject will participate in the study for approximately 3 weeks, including 2 weeks of screening, 1 week of scanning and safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Understand the study procedures and agree to participate by providing a signed informed consent form.
* Be willing and able to comply with all study procedures and restrictions.
* Be ≥ 21 years of age (a balanced gender ratio is preferred.).
* Have a body mass index (BMI) between 19-26 (inclusive).
* Be capable of laying on the scanner for a consecutive hour.
* All females of childbearing potential (premenopausal or less than 2 years post-menopausal and have not undergone surgical sterilization) must undergo a blood pregnancy test during the screening period. The results of the pregnancy test must be negative, and these participants must be using effective contraception, such as complete abstinence, condom use, IUD, etc.

Additional inclusion criteria for patients:

* Patients must have histological, pathological and/or cytological confirmation of solid malignant tumor.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* According to the investigator's judgment, the expected survival time must be more than 6 months.
* Patients must have an adequate organ function before the administration of the 68Ga-LNC1007 (in the absence of blood transfusion, hematopoietic stimulating and hepatoprotective agents), as defined by:

  1. White blood cell (WBC) count ≥ 3×109/L or absolute neutrophil count (ANC) > 1.5×109/L, platelets ≥ 100×109/L, hemoglobin (Hb) > 10.0g/dL
  2. Serum albumin > 3.0 g/dL, total bilirubin < 1.5×ULN, alanine aminotransferase (ALT) < 3×ULN, aspartate aminotransferase (AST) < 3×ULN
  3. Creatinine clearance ≥ 60 mL/min (calculated using the Cockcroft-Gault formula).

Exclusion Criteria:

* Contraindications to PET/CT scan, which include, but are not limited to, conditions like claustrophobia.
* A medical history of epilepsy or seizures, excluding febrile convulsions during childhood.
* Blood donation or otherwise major blood loss (> 400 mL) within 3 months prior to the screening or during the study period.
* Active and clinically significant bacterial, fungal, or viral infections, including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness (patients with treated HIV and hepatitis B or C could be included).
* Insufficient venous access (two different venous accesses are required for the injection of the experimental drug and PK blood sampling).
* Females who are pregnant (positive pregnancy test at screening period), lactating, or have fertility potential (premenopausal or less than 2 years post-menopausal and have not undergone surgical sterilization) and refusal to use effective contraception (such as complete abstinence, condom use, IUD, etc.) during the trial (from the signing of the informed consent form) and three months after administration.
* Males with plans for procreation or sperm donation during the trial (from the signing of the informed consent form) and three months after administration. Males who do not wish to take effective contraceptive measures should be excluded as well (such as complete abstinence, condom use, surgical sterilization, etc.).
* History of alcohol allergy, polyethylene glycol (PEG) allergy or other allergies that the investigator considers could increase the trial risk.
* Radioactive drug imaging or treatment within 7 days prior to screening.
* Participation in other clinical trials within the past 1 months before screening visit.
* Participation in clinical trials of radiopharmaceuticals within 1 year prior to screening.
* History of drug or alcohol abuse within the past year, or a long-term history of illegal drug use.
* History of long exposure to high-dose radiation.
* Other conditions that the investigator believes make the subject unsuited for participating in the trial. For example, active infections requiring intravenous antibiotic treatment 14 days prior to administration.

Additional exclusion criteria for healthy volunteers:

* Clinically significant disease or medical history as determined by the trial investigator. This includes, but is not limited to:

  1. Conditions related to circulatory, respiratory, digestive, urinary, hematological, neurological, endocrine, and musculoskeletal systems.
  2. History of mental disorders or any other disease with clinical significance.
  3. Previous major surgeries or anticipated major surgery within 1 month prior to the screening or during the study period.
* Currently having medical comorbidities that are considered to be clinically significant by investigators, such as comorbidities that may interfere with the absorption or metabolism of the investigational drug or limit the interpretation of the trial results.
* Having taken any prescription drugs, over-the-counter drugs, health products, or traditional herbal medicine within 14 days before administration.
* Abnormal findings considered clinically significant by investigators during the screening period, such as physical examination, vital signs, laboratory tests or 12-lead ECG (baseline physical examination, laboratory tests, and 12-lead ECG results are acceptable from Day -7 to Day -1).

Additional exclusion criteria for patients:

* Concurrent anti-cancer treatment.
* A history of mental disorders or any other disease with clinical significance.
* Previous major surgeries or anticipated major surgery within 1 month prior to the screening or during the study period.
* Concurrent other disease like metabolic abnormality, abnormal physical examination, or abnormal laboratory test at the time of screening, which will make the patient reasonably suspected to be unsuitable for receiving the study drug, or will affect the interpretation of the study results, or will put the subject at high risk such as idiopathic pulmonary fibrosis or lung disease, urinary incontinence, etc., according to the investigator's judgment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of 68Ga-LNC1007 Injection. | Through study completion, assessed up to 2 years
  The safety assessments of this phase I trial are based on systemic safety evaluation. The frequency and severity of Treatment emergent adverse events (TEAE) will be classified according to Common Toxicity Criteria for Adverse Events 5.0. The seriousness and relationship of study treatment will be assessed.

SECONDARY OUTCOMES:
Evaluate the radioactivity of 68Ga-LNC1007 Injection. | Through study completion, assessed up to 2 years
  Patient blood samples at 5 min, 15 min , 30 min , 60 min , 120 min , 180 min , 240 min，24 h after the administration of 68Ga-LNC1007.
  Patient urine samples at 0-1.5 h, 1.5-3 h and 3-4 h after the administration of 68Ga-LNC1007.
  All samples will be drawn for radioactivity by a gamma counter.
Evaluate the metabolites of 68Ga-LNC1007 Injection. | Through study completion, assessed up to 2 years
  Patient blood samples at 5 min , 60 min , 120 min , 180 min , 240 min，24 h after the administration of 68Ga-LNC1007.
  Patient urine samples at 0-1.5 h, 1.5-3 h and 3-4 h after the administration of 68Ga-LNC1007.
  The major metabolites will be conducted by radioHPLC.
Evaluate the radioactive counts of each target organ of 68Ga-LNC1007 Injection. | Through study completion, assessed up to 2 years
  Whole-body images will be acquired by using standard methods. The whole-body PET scan images will be evaluated and the regions of interest (ROI) such as heart, lung, liver, kidney, spleen, and brain, will be delineated on the whole-body image of each phase to obtain the radioactive counts of each target organ in each phase.
Evaluate the SUV values of 68Ga-LNC1007 Injection. | Through study completion, assessed up to 2 years
  The SUV values (SUVmax, SUVmean) of each organ will be summarized to reflect the biodistribution of 68Ga-LNC 1007 Injection in the human body.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Imaging Research Centre (CIRC) ；National University of Singapore., Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No